CLINICAL TRIAL: NCT00701532
Title: Dopamine Transporter (DAT) in Pharmacological Treatments of Cocaine Dependence. CAIMAN (Cocaine Addiction Imaging Medications and Neurotransmitters) Study
Brief Title: Brain Imaging Study of the Effects of Modafinil in Cocaine Addiction
Acronym: CAIMAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Mission Interministérielle de Lutte contre la Drogue et la Toxicomanie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P070150
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Cocaine Addiction; Cocaine Dependence
Keywords: Cocaine; Substance abuse; Addiction; Dependence; Modafinil; Brain imaging
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Behavior, Addictive | interventions — Modafinil; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Neuroimaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): active
  Interventions: Drug: Modafinil and PET (brain imaging)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Modafinil and PET (brain imaging) — duration 90 days
  Arms: 1
Drug: placebo — duration 90 days
  Arms: 2

SUMMARY:
-Context: Study objectives Primary: impact of modafinil versus placebo on DAT density modifications in the striatal and extra-striatal regions in cocaine dependent subjects hospitalised from D3 to D21.

Primary Hypothesis:

More rapid normalisation of DAT concentrations measured by PET using modafinil versus placebo from D3 to D21 during cocaine detoxification.

DETAILED DESCRIPTION:
Context:

Cocaine dependence is a disorder with a rapidly progressive evolution, associated with various complications. Because of cocaine's direct action on the dopamine transporter (DAT), dopaminergic system dysregulation plays a fundamental role in reinforcement phenomenon and in dependence. This has been proven in numerous animal and post-death human studies of striatal DAT. In vivo studies in cocaine dependent patients are rare. Currently no pharmacotherapy is available to treat this pathology. Current studies indicate that pharmacological agents such as modafinil may be able to reverse the neuroadaptations induced by cocaine dependence. However, no functional neuroimaging study (Positron Emission Tomography, PET) has analysed the impact of medications on DAT density in cocaine dependent patients. However, in primates, in vivo PET has shown modafinil affinity for DAT.

Primary Hypothesis:

More rapid normalisation of DAT concentrations measured by PET using modafinil versus placebo from D3 to D21 during therapeutic cocaine withdrawal.

Study objectives Primary: impact of modafinil versus placebo on DAT density modifications in the striatal and extra-striatal regions in cocaine dependent subjects hospitalised from D3 to D21.

Secondary:

Evaluation of the clinical efficacy of modafinil during therapeutic cocaine withdrawal. Correlation between craving measurements, depressive symptom measurements and cognitive deficit measurements observed and modifications of DAT density.

Study of DAT from D3 to D21 versus a pre-existing data base of control subjects.

Tolerance and safety evaluation of high modafinil doses, measured by adverse events and biological parameters.

Calculation of the number of subjects: A power of 90% is found for a number of subjects estimated at 24 (bilateral test, α risk at 5%, estimated SEM of 5%, variation of the occupational concentration of the DAT expected to be at least 12% in the modafinil group). Considering the usual rate of patients lost to follow-up in this patient population (25%), we plan to include 30 patients.

Methodology: This study is regulated by the law on biomedical research of August 9, 2004. It is a randomised monocentric double blind study versus placebo. During the study, for 90 days, patients will receive in double blind either modafinil or placebo according to their randomisation arm.

Evaluations will include 2 PET, cerebral MRI, blood work-up, urinary toxin screen, clinical scales for craving, depression and neuropsychological evaluations.

Patients will be recruited over 24 months. The total study length will be 36 months.

Primary judgment criteria: Variation of the linking potentials (specific fixation rate for the radioligand [11C]-PE2I to DAT) between the TEP measurement on D3 and D21 within the various anatomical region of interest between the 2 groups (modafinil, placebo).

Expected Results: Decreased DAT occupation rates in the modafinil group versus placebo from D3 to D21 of withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Men of at least 18 years of age
* Cocaine dependent according to DSM IV TR criteria
* Seeking treatment
* Capable of understanding and giving their informed written consent
* With National Health coverage
* Urinary screen positive for cocaine in the weeks prior to inclusion

Exclusion Criteria:

* Women
* Other DSM IV TR axe I diagnostic criteria (except for tobacco)
* Neurological disorders
* Treatment that interferes with the DAT and modafinil
* Contraindications for modafinil and Magnetic Resonance Imaging

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Decreased DAT occupation rates in the modafinil group versus placebo from day 3 to day of cocaine detoxification. | day 3 and day of cocaine detoxification

SECONDARY OUTCOMES:
Evaluation of the clinical efficacy of modafinil during therapeutic cocaine withdrawal. | D3 to D90
Correlation between craving measurements, depressive symptom measurements and cognitive deficit measurements observed and modifications of DAT density. | D3 to D21
Study of DAT from D3 to D21 versus a pre-existing data base of control subjects. | D3 to D21
Tolerance and safety evaluation of high modafinil doses, measured by adverse events and biological parameters. | D3 to D90

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reynaud, PhD, Study Director — Assistance Publique - Hôpitaux de Paris Hôpital Paul Brousse
Locations (2):
- France (2):
  - Unité de recherche U797 Inserm - CEA - Université Paris-Sud. " Neuroimagerie & Psychiatrie " Service Hospitalier Frédéric Joliot, Orsay
  - Centre d'Enseignement, de Recherche et de Traitements des Addictions - Hopital Universitaire Paul Brousse, Villejuif